CLINICAL TRIAL: NCT00274625
Title: Evaluation of Surgisis Gold Graft for Incision Reinforcement After Open Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Collaborators: Cook Biotech Incorporated (Industry); MED Institute, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1076-05-00; 04-007
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Results first posted 2014-11-12 (Estimated); Last update posted 2014-11-12 (Estimated); Status verified 2014-11

CONDITIONS: Hernia; Obesity
Keywords: Biomaterials; Bariatric Surgery; Hernia, Prevention of; Obesity; Bypass Surgery; Incisional Hernia; Ventral Hernia
MeSH Terms: conditions — Hernia; Obesity; Incisional Hernia; Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Surgisis Gold Graft
  Interventions: Device: Surgisis Gold Graft
- 2 (Active Comparator): Control
  Interventions: Procedure: Control

INTERVENTIONS:
Device: Surgisis Gold Graft — Surgisis Gold Graft is placed as an underlay following open bariatric surgery.
  Arms: 1
Procedure: Control — Incision is closed without the placement of a graft material (standard of care control)
  Arms: 2

SUMMARY:
The primary objective is to compare the effectiveness of the Surgisis Gold Graft to suture closure alone in preventing an incisional hernia after open bariatric surgery.

DETAILED DESCRIPTION:
This will be a prospective, randomized clinical trial comparing outcomes of use of a sublay of Surgisis Gold Graft for tissue reinforcement, as compared to suture closure alone in evaluating incidence of incisional hernias. Prior to undergoing open bariatric surgery, patients will be randomized to receive either Surgisis Gold Graft or suture closure alone. Subjects will be seen for follow-up visits at six weeks, three months, six months, one year and two years post-operatively. Patients may see their primary care physician for the one and two follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Planned operative approach via upper midline incision with goal of weight loss
* 18 years of age or older
* Body mass index (BMI) >= 30 kg/m2
* Documented history of non-surgical attempts at weight loss
* Patients undergoing reoperation for a failed previous bariatric procedure are eligible provided the operation is being performed for weight loss and provided at the time of reoperation there is no incisional hernia
* Patients with small, non-incarcerated, previously unrepaired umbilical hernias are acceptable provided the hernia defect is no greater than 2.5 cm in diameter

Exclusion Criteria:

* Patients with pre-existing midline abdominal wall incisional hernia or diastasis rectus
* Patients undergoing repeat bariatric surgery for complications of a previous bariatric procedure
* Patients with a previous upper midline incision found to have an incisional hernia
* Patients with connective tissue disorders known to predispose to hernia formation
* Active infection at the time of proposed surgery
* Sensitivity or religious objections to porcine products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2005-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sarr, MD, Principal Investigator — Mayo Clinic Foundation
Locations (2):
- United States (2):
  - Mayo Clinic Foundation, Rochester, Minnesota
  - St. Mary's Medical, Richmond, Virginia

REFERENCES:
- [Result] Sarr MG, Hutcher NE, Snyder S, Hodde J, Carmody B. A prospective, randomized, multicenter trial of Surgisis Gold, a biologic prosthetic, as a sublay reinforcement of the fascial closure after open bariatric surgery. Surgery. 2014 Oct;156(4):902-8. doi: 10.1016/j.surg.2014.06.022. PMID 25239343

RESULTS

PARTICIPANT FLOW:
Groups:
- Surgisis Gold: Surgisis Gold Graft is placed as an underlay following open bariatric surgery.
- Suture Closure: Control : Incision is closed without the placement of a graft material (standard of care control)
Period: Overall Study
Arm/Group | Surgisis Gold | Suture Closure
Started | 199 | 203
Completed | 139 | 141
Not Completed | 60 | 62
Not completed — Lost to Follow-up | 46 | 54
Not completed — Excluded from analysis | 14 | 8

BASELINE CHARACTERISTICS:
Population: 14 patients in Surgisis Gold group and 8 patients in Suture Closure group were excluded from the analysis, because prior to procedure, either they were found not to meet the inclusion/exclusion criteria, or they chose not to participate.
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgisis Gold | Suture Closure | Total
Number analyzed (Participants) | 185 | 195 | 380
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (10.6) | 45.1 (12.1) | 44.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 156 | 302
  Male | 39 | 39 | 78
Weight [Mean (Standard Deviation); unit: kg] | 138 (30) | 143 (34) | 140.6 (32.2)
BMI (Body mass index) [Mean (Standard Deviation); unit: kg/m^2] | 48.2 (8.2) | 48.2 (7.7) | 48.2 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Incisional Hernia
Description: An obvious defect or interruption of the fascia in the area of the incision that was palpable on clinical examination and/or visible by a cross-sectional imaging modality.
Time Frame: 2 years
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Surgisis Gold | Suture Closure
Number analyzed (Participants) | 185 | 195
participants | 32 | 38
Statistical Analysis 1: Comparison: Surgisis Gold vs Suture Closure; Test type: Superiority or Other; p = 0.60, Fisher Exact

ADVERSE EVENTS:
Description: 14 patients in Surgisis Gold group and 8 patients in Suture Closure group were excluded from the analysis, because prior to procedure, either they were found not to meet the inclusion/exclusion criteria, or they chose not to participate.
Arm/Group | Surgisis Gold | Suture Closure
Serious Adverse Events (participants affected / at risk) | 0/185 | 0/195
Other Adverse Events (participants affected / at risk) | 87/185 | 62/195
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgisis Gold (N=185) | Suture Closure (N=195)
Pain (General disorders) | 32 (32) | 21 (21)
Wound infection (Infections and infestations) | 23 (23) | 8 (8)
Wound erythema requiring antibiotics (Infections and infestations) | 25 (25) | 2 (2)
Incisional hernia (Infections and infestations) | 32 (32) | 38 (38)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days